CLINICAL TRIAL: NCT06762145
Title: EArly Effect of Glucocorticoid on Incidence of Persistent Left BundlE Branch Block (LBBB) Post-TAVR
Brief Title: EArly Effect of Glucocorticoid on Incidence of Persistent Left BundlE Branch Block (LBBB) Post-TAVR (EAGLE-TAVR Trial)
Acronym: EAGLE-TAVR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiao-dong Zhuang (Other)
Responsible Party: Sponsor-Investigator, Xiao-dong Zhuang, Dr., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ChiCTR 200039901; 82070384 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Transcatheter Aortic Valve Replacemen; Left Bundle Branch Block
Keywords: TAVR; LBBB; Glucocorticoid
MeSH Terms: conditions — Bundle-Branch Block | interventions — Methylprednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methylprednisolone (Experimental)
  Interventions: Drug: Methylprednisolone (Corticosteroid)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone (Corticosteroid) — Intravenous Methylprednisolone 1mg/kg/d for 3 days started from the day on TAVR
  Arms: Methylprednisolone
Drug: Placebo — Placebo for 3 days started from the day on TAVR
  Arms: Placebo

SUMMARY:
Transcatheter aortic valve replacement (TAVR) has become an established alternative for the treatment of severe symptomatic aortic stenosis irrespective of surgical risk. The development of new-onset left bundle branch block (LBBB) is the most common complication, which impairs outcomes after TAVR.

Glucocorticoid has been proven safe and effective in arrythmia after cardiac surgery. The anti-inflammatory effect of glucocorticoid may alleviate the occurrence of LBBB and thus the prognosis.

EAGLE-TAVR is a multi-center, randomized, double blind, placebo-controlled trial. A total of 200 patients selected to undergo TAVR will be randomized in a 1:1 ratio to the treatment with intravenous Methylprednisolone 1mg/kg/day or placebo for 3 days started from the day of the procedure.

According to the definition of the Valve Academic Research Consortium 3, persistent LBBB is defined as present LBBB at discharge or >7 days post-TAVR. The primary endpoint is the occurrence of new-onset LBBB at 30 days post TAVR.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years
2. Selected to undergo transfemoral TAVR based on heart team decision

Exclusion Criteria:

1. Allergic to Methylprednisolone
2. Patients with a prior pacemaker or high degree atrioventricular block
3. Septicemia
4. Life expectancy < 1 year irrespective of heart disease (Cancer, severe liver disease, severe renal disease, severe pulmonary, et al)
5. Inability to provide written informed consent
6. Participation in another clinical trial with an active intervention
7. Patients on prior chronic treatment with glucocorticoids (both oral, inhaled, or intravenous, but topical and ophthalmic administration is allowed)
8. Gastrointestinal bleeding
9. Acute myocardial infarction within 1 month
10. Intracardiac thrombus or vegetation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of persistent LBBB | 30 days
  Assessed based on electrocardiogram performed at admission, every day post TAVR until discharge. New-onset LBBB is defined as LBBB with no RBBB before the procedure and high degree atrioventricular block with RBBB before the procedure. Persistent LBBB is defined as present LBBB at discharge or >7 days post-TAVR.

SECONDARY OUTCOMES:
Occurrence of permanent LBBB | 1 year
  Present LBBB >30 days post-TAVR
Occurrence of syncope | 30 days and 1 year
  Assessed based on symptoms
Incidence of permanent pacemaker implantation | 30 days and 1 year
  Assessed based on operation history
Rehospitalization rate | 30 days and 1 year
  According to medical history or telephone follow-ups
The changes of left ventricular ejection fraction | 30 days and 1 year
  Evaluated based on echocardiogram
The incidences of major clinical adverse events | 30 days and 1 year
  All-cause mortality, cardiovascular mortality, stroke, myocardial infarction

OTHER OUTCOMES:
Safety Outcome | 30 days and 1 year
  Incidence of clinically severe side effects possibly related to study drug intake like infection, gastrointestinal bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No